CLINICAL TRIAL: NCT01113034
Title: A Phase 1 Randomized Double-Blind Placebo-Crossover Safety Trial of DAS181 (Fludase®) in Adult Subjects With Well-Controlled Asthma or Bronchiectasis
Brief Title: A Safety Trial of DAS181 (Fludase®) in Adult Subjects With Well-Controlled Asthma or Bronchiectasis
Acronym: DAS181
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAS181 - 1 - 04, 10 - I - 0085; NCT01131286 (obsolete NCT alias)
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2010-07

CONDITIONS: Asthma; Bronchiectasis
Keywords: Asthma; Bronchiectasis
MeSH Terms: conditions — Asthma; Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAS181 Dry Powder 10 mg qd x 3 days (Active Comparator)
  Interventions: Drug: DAS181 dry powder, formulation F02
- Lactose Placebo (Placebo Comparator)
  Interventions: Drug: Respitose ML006 (DMV-Fonterra)

INTERVENTIONS:
Drug: DAS181 dry powder, formulation F02 — 10 mg delivered dose DAS181 in clear HPMC #3 Capsules
  Arms: DAS181 Dry Powder 10 mg qd x 3 days
Drug: Respitose ML006 (DMV-Fonterra) — Lactose monohydrate
  Arms: Lactose Placebo

SUMMARY:
The primary objective is to evaluate whether DAS181 is safe in subjects with well-controlled asthma or bronchiectasis.

DETAILED DESCRIPTION:
This study will assess the safety of a new study drug called DAS181 (Fludase®). This study is being done with NexBio, Inc., the company that makes DAS181 (Fludase®). DAS181 is not approved by the Food and Drug Administration (FDA); however the FDA has given permission to use DAS181 in human studies. To date, DAS181 has been given to about 81 healthy people and has been well tolerated with no reported serious adverse reactions. This is the first experimental study to test if it is safe to use this drug in people with well-controlled asthma or bronchiectasis. DAS181 is not being given to treat asthma or bronchiectasis, but to learn if it is safe to use in people with well-controlled asthma or bronchiectasis. DAS181 is being developed as a medication to prevent and treat infections due to common respiratory viruses like influenza (including the pandemic H1N1 strain), parainfluenza, and other viruses. New drugs to treat respiratory viruses are needed because some currently available drugs are not effective against some types or strains of viruses. Drugs that are effective against respiratory viruses are especially important for people with asthma or bronchiectasis because these lung conditions increase the risk of serious complications due to respiratory virus infections. Making sure the new drug is safe in people with asthma or bronchiectasis is important because people with these lung conditions may have different side effects from a drug than people who don't have asthma or bronchiectasis. We plan to enroll 24 volunteers into the study: 12 persons with well-controlled asthma and 12 persons with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female subject must be 18 to 65 years of age.
2. Except for underlying airway disease, subject must be in good health as determined by medical history, targeted physical examination based on medical history, and vital signs (that include temperature, blood pressure, heart rate, and pulse oximetry).
3. Subject must be able to verbalize understanding of the informed consent form, verbalize willingness to complete all study procedures, and provide written informed consent (sign the informed consent form).
4. Subject must be willing to commit to participating in both the initial and cross-over stages of the study.
5. Dipstick analysis of subject's urine specimen must be negative or show only trace amounts of glucose, hemoglobin, and protein. A menstruating female who tests positive for urine hemoglobin may be retested.
6. Subject must have blood screening test results that are within normal limits (according to standards set within the Clinical Center) for the following tests: alanine transaminase (ALT), alkaline phosphatase (ALKP), activated partial thromboplastin time (APTT), and aspartate transaminase (AST).
7. Subject must have hematologic screening tests that are within a specified range, including hemoglobin of 10.9 g/dL, white blood cell count 2500/mm3, and platelet count 125,000/mm3 (all <grade 1 on DAIDS severity scale).
8. A female subject must be post-menopausal (1 year without menses), have been surgically sterilized, practice abstinence, or use an effective method of birth control that may include an intrauterine device, spermicide, barrier, and hormonal contraception. A female subject must also have a negative serum test for pregnancy during the Screening period, and a negative urine test for pregnancy on the first day of drug or placebo administration.

Asthma Subjects:

1. Subject must have a clinically established diagnosis of asthma based upon a history of episodic symptoms of airway obstruction or airway hyper-responsiveness (i.e., wheezing).
2. Subject must have a documented increase in FEV1 or forced vital capacity (FVC) 12% (and at least 200 mL) from baseline after inhaling a short-acting bronchodilator; or a PC20FEV1 response to methacholine (i.e., the concentration of methacholine that produces a 20% decrease in FEV1 from the post-saline value during the methacholine challenge) of 8 mg/mL.
3. At the time of study enrollment, subject's asthma has been well-controlled for at least the past 3 months, as defined by the following:

   1. Daytime symptoms occur 2 days per week
   2. Normal daily activity is not limited by asthma
   3. Nocturnal symptoms/nighttime awakenings 2 times/month
   4. FEV1 80% predicted
   5. Use of short-acting beta-agonist 2 days/week
   6. Exacerbations requiring oral corticosteroids occur 2 times/year
   7. There has been no change in asthma medication dose or regimen within 3 months of study enrollment
   8. Not currently taking oral corticosteroids

Bronchiectasis Subjects:

1. Subject will be recruited from ongoing NIH natural history protocols (06-I-0217, 01-I-0202, and 09-I-0172) and/or the National Bronchiectasis Registry.
2. Subject must have a pre-established diagnosis of bronchiectasis based on chest computed tomography (CT) scan findings within 12 months of enrollment (no diagnostic CT scans will be performed during the Screening phase of this study).
3. Subject must not have overt allergic bronchopulmonary aspergillosis, cystic fibrosis, or primary ciliary dyskinesia.
4. Subject's bronchiectasis is stable as defined by the following:

   a. Less than 2 acute exacerbations in the preceding 12 months and none in the preceding 4 weeks, with acute exacerbation defined as persistent (>24 hour) worsening of >3 respiratory symptoms associated with bacterial infection including: i. Cough ii. Dyspnea iii. Hemoptysis iv. Increased sputum purulence or volume v. Chest pain b. No change in antimicrobial regimen for at least 3 months before enrollment c. FEV1 80% predicted d. Use of short-acting beta-agonist 2 days/week for at least the past 3 months e. No baseline requirement for oxygen supplementation f. Ability to maintain oxyhemoglobin saturation of 90% during and after 6-minute walk test g. Not currently taking oral corticosteroids

Exclusion Criteria:

1. Subject has received any investigational drug or vaccine within 4 weeks prior to study drug dosing, or is planning to participate in another investigational drug or vaccine trial prior to completion of this study.
2. Subject is currently taking theophylline or oral corticosteroids.
3. Subject is allergic to milk or milk products.
4. Subject currently smokes tobacco or has smoked tobacco within 1 year prior to study enrollment.
5. Subject has a baseline requirement for oxygen supplementation.
6. Subject is unable to maintain an oxyhemoglobin saturation of 90% during and after 6-minute walk test.
7. The subject tests positive for human immunodeficiency virus (HIV), for hepatitis B virus (HBV), or hepatitis C virus (HCV).
8. The subject's resting blood pressure is outside normal limits (defined as: systolic 90-140 mmHg; diastolic 50-90 mm Hg).
9. The subject's heart rate is less than 45 or greater than 100 beats per minute at rest.
10. The subject weighs less than 45 kg.
11. The subject has a Body Mass Index of greater than 35 kg/m2.
12. The subject has experienced an episode of acute upper respiratory tract infection, pneumonia, otitis, bronchitis, or sinusitis within 6 weeks of study enrollment.
13. The subject has an oral temperature above 37.8°C (100°F).
14. The subject has any surgical, medical, or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism, or excretion of the drug.
15. The subject has overt primary ciliary dyskinesia, allergic bronchopulmonary aspergillosis, or cystic fibrosis.
16. The subject has previous or current history of the following conditions: renal, hepatic, cardiac, hematologic (including sickle cell disease), muscular, neurological, metabolic, or immunological disorders, malignancy, hepatitis or cirrhosis, transplant recipients, HIV-infection, or other immunosuppressive illness, which could, in the opinion of the study investigators, compromise subject safety or interfere with the assessment of study drug safety.
17. A female who is pregnant or breast-feeding.
18. A subject who has received blood products within 6 months of study enrollment.
19. The subject has donated or lost more than 500 mL of blood in the 3 months prior to screening.
20. The subject has clinically significant medical or psychological conditions that would compromise the subject's safety, influence the results of the study, affect the subject's ability to participate in the study, or impair the subject's ability to provide informed consent.
21. The subject has a history of alcoholism, drug dependence, or significant psychiatric illness within 2 years of study enrollment.
22. The subject uses anticoagulant medications or drugs with known potential for hepatotoxicity as such agents could interfere with relevant safety assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08-22 (Actual); Study Completion 2011-08-22 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity profile: Unacceptable Serious Adverse Events | 6 weeks (up to 12 weeks)

SECONDARY OUTCOMES:
Assessment of acute tolerability of DAS181 administration in subjects with well-controlled asthma or bronchiectasis, specifically with regard to airway obstruction (FEV1) and oxyhemoglobin saturation. | 6 weeks
Examine potential effects of DAS181 on underlying lung disease, i.e., as relates to airway hyperreactivity, mucus production, airway inflammation, frequency of acute exacerbations, and health related quality of life measurements. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Moss, MD, Study Director — Ansun Biopharma, Inc.; Kenneth Olivier, MD, MPH, LCID, NIAID, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- NIH Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Davey EL, Colombo RE, Fiorentino C, Fahle G, Davey RT Jr, Olivier KN, Kovacs JA. Pneumocystis colonization in asthmatic patients not receiving oral corticosteroid therapy. J Investig Med. 2017 Apr;65(4):800-802. doi: 10.1136/jim-2016-000381. Epub 2017 Feb 13. PMID 28193704
- [Derived] Colombo RE, Fiorentino C, Dodd LE, Hunsberger S, Haney C, Barrett K, Nabha L, Davey RT Jr, Olivier KN. A phase 1 randomized, double-blind, placebo-controlled, crossover trial of DAS181 (Fludase(R)) in adult subjects with well-controlled asthma. BMC Infect Dis. 2016 Feb 1;16:54. doi: 10.1186/s12879-016-1358-9. PMID 26830468